CLINICAL TRIAL: NCT06841952
Title: A Prospective, Two-arm, Multi-center Clinical Study of the Efficacy and Safety of Tretinoin Capsules Combined With Azacitidine and Venetoclax in Treatment Naïve Participants With Acute Myeloid Leukemia
Brief Title: Study of Tretinoin Capsules in Combination With Azacitidine and Venetoclax in Treatment Naïve Participants With Acute Myeloid Leukemia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Responsible Party: Principal Investigator, HAN Yue, Chief of Service, The First Affiliated Hospital of Soochow University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: SOOCHOW-HY-2024-12-10
Record Dates: First submitted 2025-01-15; First posted 2025-02-24 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: AML, Adult
Keywords: tretinoin; azacitidine; venetoclax
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ATRA+VEN+AZA arm (Experimental): (1)Inductive therapy: AZA 75mg/m² per day for days 1-7 and venetoclax 100mg orally for day 1 , 200mg orally for day 2, 300mg orally for day3-5, 400mg orally for day6-9,ATRA capsule 45mg/m² orally for day 11-28, every 28 days for 2 cycles or progression; (2)Consolidate therapy:AZA 75mg/m² per day for days 1-7 and venetoclax 100mg orally for day 1 , 200mg orally for day 2, 300mg orally for day3-5, 400mg orally for day6-9,ATRA capsule 45mg/m² orally for day 11-28, every 28 days for 2 cycles or progression; (3) Maintenance therapy:ATRA 45mg/m2 orally for d1-21 every 28 days,AZA 75mg/m² per day for days 1-7.Maintenance treatment was given once a month for 4 times, then once every 3 months until progression.
  After the second induction therapy, allogeneic hematopoietic stem cell transplantation was recommended for patients with suitable donors.
  Interventions: Drug: ATRA+Venetoclax+Azacitidine
- DNR+ Ara-C arm (Active Comparator): (1)Inductive therapy: Daunorubicin 60mg/m² d1-3，cytarabine100mg/m² d1-7, every 28 days for 2 cycles or progression; (2)Consolidate therapy:Intermediate-dose cytarabine alone or combined with anthracyclines is recommended (cytarabine 1.5-2g/m²), every 28 days for 2 cycles or till progression. (3) Maintenance therapy:AZA 75mg/m² per day for days 1-7 every 28 days.Maintenance treatment was given once a month for 4 times, then once every 3 months until progression.
  After the second induction therapy, allogeneic hematopoietic stem cell transplantation was recommended for patients with suitable donors.
  Interventions: Drug: Chemotherapy drug

INTERVENTIONS:
Drug: ATRA+Venetoclax+Azacitidine — Participants will receive a standard dose of azacitidine (75mg/m²/day)，venetoclax (target dose, 400 mg)，ATRA 45mg/m²/day
  Arms: ATRA+VEN+AZA arm
Drug: Chemotherapy drug — Participants will receive commercially available cytarabine (cytosine arabinoside) and anthracycline (daunorubicin).
  Arms: DNR+ Ara-C arm

SUMMARY:
This study was a prospective, two-arm, multicenter clinical trial to evaluate the efficacy and safety of tretinoin capsules combined with azacitidine and venetoclax in the treatment of newly diagnosed acute myeloid leukemia. Azacitidine, venetoclax, and tretinoin may arrest cancer cell growth by demethylation, promoting cell differentiation, or killing cells, while reducing blood-related adverse effects by promoting cell differentiation.

DETAILED DESCRIPTION:
This is a multi-center, non-controlled, open-label, Phase 3 interventional study.Young (≥18 and ≤60 years old) patients with newly diagnosed non M3, acute myeloid leukemia will receive a combination of AZA+Venetoclax+ATRA(AVA regimen) or daunorubicin +cytarabine(DA regimen) as induction treatment for 2 cycles.

According to standard procedures, patients will receive one of the following consolidation regimens separately, including the AVA regimen, or medium-dose cytarabine alone or in combination with anthracyclines regimen for 2cycle. After consolidation therapy, maintenance treatment could be given once a month for 4 times, then once every 3 months until progression.

After the second induction therapy, allogeneic hematopoietic stem cell transplantation was recommended for patients with suitable donors.

The primary endpoint is ORR after second induction therapy.Outcome measures included complete remission (CR)/complete remission with incomplete hematologic recovery (CRi) .

ELIGIBILITY:
Inclusion Criteria:

* Patients initially diagnosed with AML (excluding APL) according to WHO diagnostic criteria.
* Patients who have not previously received other induction therapies (excluding hydroxyurea and leukapheresis).
* Total white blood cell (WBC) count ≤ 25 × 10^9/L.
* Ages 18 to 60 years, inclusive, with no gender restrictions.
* ECOG Performance Status score of 0-2.
* Total bilirubin ≤ 3 times the upper limit of normal (ULN); Alanine aminotransferase (ALT) ≤ 3 times ULN; Aspartate aminotransferase (AST) ≤ 3 times ULN; (excluding leukemia infiltration).
* Endogenous creatinine clearance rate ≥ 30 ml/min.
* Enrolled patients must be capable of understanding and willing to participate in the study, and must sign the informed consent form.

Exclusion Criteria:

* Patients with Acute Promyelocytic Leukemia (APL).
* Patients with concomitant central nervous system leukemia or extramedullary leukemia involvement, such as testicular infiltration.
* Patients with current or historical immunodeficiency virus infection.
* Patients with active Hepatitis B or Hepatitis C infection.
* Patients with a history of drug allergy, including but not limited to etoposide, azacitidine, venetoclax, daunorubicin, and cytarabine.
* Patients with active or progressive malignant tumors or severe infections.
* Patients with a left ventricular ejection fraction (LVEF) of less than 30%, classified as New York Heart Association (NYHA) Class III or above, and those deemed ineligible for enrollment by the investigator.
* Patients who are pregnant or breastfeeding.
* Patients who refuse to participate in the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 158 (Estimated)
Dates: Start 2025-02-15 (Estimated); Primary Completion 2028-12-15 (Estimated); Study Completion 2030-12-15 (Estimated)

PRIMARY OUTCOMES:
The overall response rate (ORR) after the second therapy | Efficacy was assessed within 2 weeks after completion of the second course of therapy or within 1 week before the third course of therapy
  ORR rate was defifined as patients achieving a CRc or PR
The composite complete remission rate (CRc) after the second therapy | Efficacy was assessed within 2 weeks after completion of the second course of therapy or within 1 week before the third course of therapy
  complete response (CR) plus complete response with incomplete blood count recovery (CRi)] after 2 cycles of treatment.

SECONDARY OUTCOMES:
Composite complete response (CRc) after the first therapy | Efficacy was assessed within 2 weeks after completion of the first course of induction therapy or within 1 week before the second course of therapy
  CRc rate was defifined as patients achieving a CR or CRi
The overall response rate (ORR) after the first therapy | Efficacy was assessed within 2 weeks after completion of the first course of induction therapy or within 1 week before the second course of therapy
  ORR rate was defifined as patients achieving a CRc or PR
Rate of transfusion independence | Up to 28 days after the start of therapy
  Rate of transfusion independence (TI) , including platelet transfusion independence rate and red blood cell transfusion independence rate.
Overall Survival (OS) | up to 2 years after the date of the last enrolled participants
  (OS) refers to the length of time from randomization until the death of the patient from any cause.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2025-02-02): https://cdn.clinicaltrials.gov/large-docs/52/NCT06841952/Prot_000.pdf